CLINICAL TRIAL: NCT00938392
Title: Immunogenicity and Safety Study of GSK Biologicals' Influenza Vaccine GSK2186877A in Elderly Adults.
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Investigational Influenza Vaccine for the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112662
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2186877A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- FluNG Aged Group (Experimental): Subjects receiving 1 dose of an aged lot of FLU NG vaccine (GSK2186877A).
  Interventions: Biological: GSK investigational FluNG vaccine GSK2186877A, aged lot
- FluNG Fresh Group (Experimental): Subjects receiving 1 dose of a fresh lot of FLU NG vaccine (GSK2186877A).
  Interventions: Biological: GSK investigational FluNG vaccine GSK2186877A, fresh lot

INTERVENTIONS:
Biological: GSK investigational FluNG vaccine GSK2186877A, aged lot — Single dose, intramuscular injection
  Arms: FluNG Aged Group
Biological: GSK investigational FluNG vaccine GSK2186877A, fresh lot — Single dose, intramuscular injection
  Arms: FluNG Fresh Group

SUMMARY:
The objective of the study is to evaluate immunogenicity between different formulations of GSK Biologicals' investigational vaccine GSK2186877A.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study. Specific attention should be given to the compliance potential of subjects with suspected or known drug or alcohol abuse.
* A man or woman 65 years of age or older at the time of vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation before entering into the study.

Exclusion Criteria:

* Any confirmed or suspected influenza illness within the last 6 months.
* Previous vaccination against influenza with any seasonal vaccine since December 2008.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to Visit 2.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone >= 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s) including egg and chicken protein, included history of hypersensitivity to a previous dose of influenza vaccine.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature >= 37.5°C on oral setting.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Any medical conditions in which intramuscular injections are contraindicated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 726 (Actual)
Dates: Start 2009-07-30; Primary Completion 2009-10-05 (Actual); Study Completion 2009-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Veľký Biel

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects enrolled in the study did not receive any vaccination, and as such are not accounted for as started.
Period: Overall Study
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Started | 362 | 362
Completed | 360 | 358
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluNG Aged Group | FluNG Fresh Group | Total
Number analyzed (Participants) | 362 | 362 | 724
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (6.09) | 73.5 (6.36) | 73.4 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 243 | 482
  Male | 123 | 119 | 242

OUTCOME MEASURES:

1. Primary Outcome: Serum Haemagglutination-Inhibition (HI) Antibody Titers Against the 3 Vaccine Strains
Description: Titers are presented as Geometric Mean Titers. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity including all evaluable subjects for whom data concerning immunogenicity outcome variable measures were available for the specific time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 357 | 355
Titer
  A/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  A/Brisbane [Day 0] | 14.1 [12.7 to 15.8] | 13.4 [12.1 to 14.9]
  A/Brisbane [Day 21]: number analyzed (Participants) | 357 | 354
  A/Brisbane [Day 21] | 108.4 [95.8 to 122.6] | 108.7 [95.1 to 124.1]
  A/Uruguay [Day 0]: number analyzed (Participants) | 356 | 355
  A/Uruguay [Day 0] | 18.5 [16.1 to 21.3] | 19.1 [16.7 to 21.8]
  A/Uruguay [Day 21] | 291.5 [251.9 to 337.4] | 282.7 [244.6 to 326.8]
  B/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  B/Brisbane [Day 0] | 68.2 [59.3 to 78.4] | 62.3 [54.8 to 70.7]
  B/Brisbane [Day 21] | 537.9 [483.6 to 598.3] | 534.2 [483.5 to 590.3]

2. Secondary Outcome: Number of Subjects Seropositive Against the 3 Vaccine Strains
Description: A seropositive subject was defined as a subject with a serum HI titer greater than or equal to 1:10. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 357 | 355
Participants
  A/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  A/Brisbane [Day 0] | 224 | 220
  A/Brisbane [Day 21]: number analyzed (Participants) | 357 | 354
  A/Brisbane [Day 21] | 353 | 349
  A/Uruguay [Day 0]: number analyzed (Participants) | 356 | 355
  A/Uruguay [Day 0] | 231 | 236
  A/Uruguay [Day 21] | 353 | 353
  B/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  B/Brisbane [Day 0] | 326 | 335
  B/Brisbane [Day 21] | 357 | 355

3. Secondary Outcome: Number of Subjects Seroconverted for the 3 Vaccine Strains
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a four-fold increase in post-vaccination titer. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane.
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity including all evaluable subjects for whom data concerning immunogenicity outcome variable measures were available for the specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 356 | 355
Participants
  A/Brisbane: number analyzed (Participants) | 356 | 354
  A/Brisbane | 228 | 227
  A/Uruguay | 292 | 292
  B/Brisbane | 224 | 247

4. Secondary Outcome: Seroconversion Factor for the 3 Vaccine Strains
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane.
Time Frame: At Day 21
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 356 | 355
Fold Increase
  A/Brisbane: number analyzed (Participants) | 356 | 354
  A/Brisbane | 7.7 [6.6 to 8.9] | 8.1 [6.9 to 9.5]
  A/Uruguay | 15.8 [13.4 to 18.6] | 14.8 [12.7 to 17.3]
  B/Brisbane | 7.9 [6.8 to 9.3] | 8.6 [7.4 to 9.9]

5. Secondary Outcome: Number of Subjects Seroprotected for the 3 Vaccine Strains
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 357 | 355
Participants
  A/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  A/Brisbane [Day 0] | 87 | 85
  A/Brisbane [Day 21]: number analyzed (Participants) | 357 | 354
  A/Brisbane [Day 21] | 318 | 308
  A/Uruguay [Day 0]: number analyzed (Participants) | 356 | 355
  A/Uruguay [Day 0] | 120 | 131
  A/Uruguay [Day 21] | 338 | 337
  B/Brisbane [Day 0]: number analyzed (Participants) | 356 | 355
  B/Brisbane [Day 0] | 261 | 260
  B/Brisbane [Day 21] | 357 | 355

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms and Any, Grade 3 and Related Solicited General Symptoms
Description: Local symptoms assessed include ecchymosis, pain, redness and swelling. General symptoms assessed include arthralgia, fatigue, gastrointestinal symptoms, headache, muscle aches, shivering and fever [oral temperature greater than or equal to 38 degrees Celsius (°C)]. Grade 3 pain: considerable pain at rest, which prevented normal everyday activities. Grade 3 ecchymosis, redness and swelling: more than 100 millimeter. Grade 3 fever: oral temperature greater than or equal to 39°C. Related: general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort including all vaccinated subjects with their symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 360 | 360
Participants
  Any Ecchymosis | 9 | 11
  Grade 3 Ecchymosis | 0 | 0
  Any Pain | 180 | 190
  Grade 3 Pain | 0 | 2
  Any Redness | 99 | 106
  Grade 3 Redness | 0 | 2
  Any Swelling | 45 | 69
  Grade 3 Swelling | 0 | 2
  Any Arthralgia | 49 | 63
  Grade 3 Arthralgia | 2 | 0
  Related Arthralgia | 28 | 44
  Any Fatigue | 86 | 98
  Grade 3 Fatigue | 1 | 1
  Related Fatigue | 68 | 80
  Any Gastrointestinal symptoms | 29 | 29
  Grade 3 Gastrointestinal symptoms | 0 | 1
  Related Gastrointestinal symptoms | 17 | 15
  Any Headache | 66 | 82
  Grade 3 Headache | 0 | 0
  Related Headache | 47 | 62
  Any Muscle aches | 60 | 62
  Grade 3 Muscle aches | 2 | 1
  Related Muscle aches | 47 | 49
  Any Shivering | 28 | 26
  Grade 3 Shivering | 2 | 0
  Related Shivering | 20 | 23
  Any Fever | 6 | 9
  Grade 3 Fever | 1 | 1
  Related Fever | 4 | 9

7. Secondary Outcome: Duration of Solicited Local and General Symptoms
Description: Local symptoms assessed include ecchymosis, pain, redness and swelling. General symptoms assessed include arthralgia, fatigue, gastrointestinal symptoms, headache, muscle aches, shivering and fever. Duration is expressed as median number of days the specific symptom was experienced.
Time Frame: During the 7-day post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, on those subjects reporting the specific symptom only.
Measure: Median (Full Range); unit: Days
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 180 | 190
Days
  Ecchymosis: number analyzed (Participants) | 8 | 11
  Ecchymosis | 4.0 [1.0 to 6.0] | 4.0 [1.0 to 7.0]
  Pain | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Redness: number analyzed (Participants) | 99 | 106
  Redness | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Swelling: number analyzed (Participants) | 45 | 69
  Swelling | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0]
  Arthralgia: number analyzed (Participants) | 49 | 63
  Arthralgia | 4.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Fatigue: number analyzed (Participants) | 86 | 98
  Fatigue | 2.5 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 28 | 29
  Gastrointestinal symptoms | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache: number analyzed (Participants) | 66 | 82
  Headache | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Muscle aches: number analyzed (Participants) | 60 | 62
  Muscle aches | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Shivering: number analyzed (Participants) | 27 | 26
  Shivering | 1.0 [1.0 to 4.0] | 1.5 [1.0 to 5.0]
  Fever: number analyzed (Participants) | 4 | 9
  Fever | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 21-day post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort including all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 362 | 362
Participants
  Any AEs | 13 | 24
  Grade 3 AEs | 1 | 1
  Related AEs | 5 | 12

9. Secondary Outcome: Number of Subjects Reporting Adverse Events of Specific Interest (AESI)
Description: AESIs for safety monitoring included autoimmune diseases and other immune mediated inflammatory disorders.
Time Frame: During the 21-day post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort including all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 362 | 362
Participants | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (up to Day 21)
Population: The analysis was performed on the Total Vaccinated Cohort including all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Number analyzed (Participants) | 362 | 362
Participants
  Any SAEs | 1 | 1
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were reported during the entire study (up to Day 21). Other Frequent (non-serious) Adverse Events were reported during a 7-day follow-up period after vaccination.
Description: Systematically assessed Other Frequent (non-serious) adverse events were reported for subjects with a completed symptom sheet only.
Arm/Group | FluNG Aged Group | FluNG Fresh Group
Serious Adverse Events (participants affected / at risk) | 1/362 | 1/362
Other Adverse Events (participants affected / at risk) | 242/362 | 252/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluNG Aged Group (N=362) | FluNG Fresh Group (N=362)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FluNG Aged Group (N=362) | FluNG Fresh Group (N=362)
Pain at the injection site (General disorders) | 180 | 190
Redness at the injection site (General disorders) | 99 | 106
Swelling at the injection site (General disorders) | 45 | 69
Arthralgia (General disorders) | 49 | 63
Fatigue (General disorders) | 86 | 98
Gastrointestinal symptoms (General disorders) | 29 | 29
Headache (General disorders) | 66 | 82
Muscle aches (General disorders) | 60 | 62
Shivering (General disorders) | 28 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.